CLINICAL TRIAL: NCT03330639
Title: The Role of Topical Capsaicin in Treatment of Rhinogenic Headache
Brief Title: Capsaicin in Treatment of Rhinogenic Headache
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant funding for study was not obtained.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0511-17-FB
Record Dates: First submitted 2017-07-27; First posted 2017-11-06 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Headache Disorders
MeSH Terms: conditions — Headache Disorders | interventions — Capsaicin

STUDY DESIGN:
Intervention Model Description: Randomized parallel group
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): This group will receive the capsaicin. The Study Drug ICX72 or sinus buster which is a homeopathic blend of capsicum annum and eucalyptol, that is readily available over the counter.
  Interventions: Other: Capsaicin
- Placebo Group (Placebo Comparator): This group will receive saline. The Placebo formulation contained saline and eucalyptol in a concentration that matched the control.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Capsaicin — Capsaicin is a homeopathic medication and there for this drug is not subject to the requirements of the FDA.
  Arms: Experimental Group
Other: Placebo — This group will receive the saline placebo solution.
  Arms: Placebo Group

SUMMARY:
Description: Capsaicin (8- methyl-N-vanillyl-6-nonenamide) has been demonstrated to have a therapeutic effect in idiopathic rhinitis. We hypothesize that capsaicin has a therapeutic effect on rhinogenic headaches, in addition to the previously studied decongestive effects. This study aims to evaluate capsaicin impact on headaches attributed to V1, V2 distribution of the sinonasal cavity. This study is a randomized, double-blinded, parallel trial.

DETAILED DESCRIPTION:
1. Title: The role of capsaicin in treatment of rhinogenic headache
2. Description: Capsaicin (8- methyl-N-vanillyl-6-nonenamide) has been demonstrated to have a therapeutic effect in idiopathic rhinitis, migraines and cluster headaches. We hypothesize that capsaicin has a therapeutic effect on rhinogenic headaches as well. This study aims to evaluate capsaicin impact on headaches attributed to the nose and paranasal sinus distribution.
3. Interventions, evaluations, and follow-up: Subjects are recruited from an Otolaryngology clinic, where a formal headache questionnaire is administered in-office, and standard endoscopy is performed in office to rule out confounding causes of headache and sinonasal disease. Written instructions are provided and consent obtained. A symptom journal is provided. Subjects are randomly selected to receive two bottles of either eucalyptol spray (placebo) or sinus buster (capsaicin) spray and are blinded to the content of the spray bottle. They are instructed to use the nasal spray one to two times daily. Subjects are permitted to continue to take headache medication as needed, but it must be recorded in their symptom journal. The journal is completed daily, and includes medication use, a headache pain score, and side effect log. Additionally, subjects fill out SinoNasal Outcome test (SNOT)22 at 2 weeks, 4 weeks, and 8 weeks. Weekly emails are sent to remind subject to fill out their journal. A phone call is made to the subject to survey them on progress at 2 and 6 weeks. Follow up visits are scheduled at 4 weeks and 8 weeks, or sooner if problems arise. A standard nasal endoscopy is performed at the first and last visit.
4. Additional data that would be tracked: Quality of life score as measured by SNOT-22 scores, treatment failure and drop-outs, and objective changes in sinus endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Consenting Adults aged 19-100 presenting to the Otolaryngology DepartmentofUniversityof Nebraska Medical center complaining of headaches/ facial pain and pressure Diagnosis of a primary rhinogenic headache disorder by the senior authors.

Exclusion Criteria:

* Exclusion criteria include: pregnancy, age less than 19, active history of smoking, presence of confirmed sinonasal disease, fibromyalgia, poorly controlled chronic health problems, allergies to chili peppers or any ingredient in the nasal spray, or confirmed Temporal Mandibular Joint (TMJ) arthralgia as the etiology of primary headache.

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
headache medication use | 1 year
  We will track the amount of headache medication used during the study period

SECONDARY OUTCOMES:
number of patients with treatment related adverse events | 1 year
  patients will be asked to report any adverse reactions or events during the study period.
headache frequency and severity | 1 year
  Patient will be asked to record the number of headaches during the study period, and record the severity from 1-10 on the Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Christie Barnes, MD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gevorgyan A, Segboer C, Gorissen R, van Drunen CM, Fokkens W. Capsaicin for non-allergic rhinitis. Cochrane Database Syst Rev. 2015 Jul 14;2015(7):CD010591. doi: 10.1002/14651858.CD010591.pub2. PMID 26171907